CLINICAL TRIAL: NCT07272993
Title: The Effect of Golden Rice Cookies With Piper Crocatum on the Prevention of Diabetic Neuropathy in Patients With Diabetes Mellitus
Brief Title: Effect of Golden Rice-Piper Crocatum Cookies on Neuropathy Prevention in Diabetes
Acronym: GRIP-DN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Herlina Husen, S.Kep.,Ns, Hasanuddin University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UH2508103
Record Dates: First submitted 2025-09-30; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Neuropathy; Diabetes Mellitus (DM); Functional Food; Nutritional Intervention; Blood Glucose
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized controlled trial using a pre-test and post-test design with a control group. Eligible participants are patients diagnosed with diabetes mellitus who present with symptoms of diabetic neuropathy. Participants will be randomly assigned into two groups: the intervention group receiving golden rice cookies enriched with Piper crocatum extract, and the control group receiving golden rice cookies without Piper crocatum.
  The intervention will be administered for 28 consecutive days, with both groups monitored under similar conditions. Assessments will be conducted at baseline (pre-test) and after the intervention period (post-test). The primary outcome measure is the change in Neuropathy Symptom Score (NSS), while secondary outcomes include blood glucose monitoring and simple neuropathy screening tests (monofilament test).
  This interventional model allows for direct comparison between the functional food intervention and the control to determine the ef
Who Masked: Participant
Masking Description: In this study, participants will not be informed whether they are receiving golden rice cookies with Piper crocatum extract or golden rice cookies without Piper crocatum. The cookies are prepared to be similar in appearance, texture, and packaging to minimize bias. Outcome assessors who evaluate neuropathy symptoms using the Neuropathy Symptom Score (NSS) and perform the monofilament test will also be masked to group assignment.
  This masking strategy is intended to reduce reporting bias from participants and measurement bias from outcome assessors, ensuring the reliability of the study results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Golden Rice Cookies Enriched with Piper Crocatum (Experimental): Participants assigned to this arm will receive cookies formulated with golden rice flour and enriched with Piper crocatum (red betel leaf extract). The cookies are consumed daily over a 28-day period. This intervention is designed to evaluate the potential neuroprotective effects of Piper crocatum in preventing or reducing symptoms of diabetic neuropathy among patients with type 2 diabetes mellitus. The formulation aims to leverage the antioxidant and anti-inflammatory properties of Piper crocatum in combination with the nutritional benefits of golden rice
  Interventions: Dietary Supplement: Golden Rice Cookies With Piper Crocatum
- Golden Rice Cookies Without Piper Crocatum (Active Comparator): Participants in this arm will receive cookies made exclusively from golden rice flour, without the addition of Piper crocatum. These cookies are also consumed daily for 28 days. This control intervention is intended to isolate the effect of Piper crocatum by comparing outcomes with the experimental group. Both cookie types are matched in appearance, taste, and packaging to maintain blinding integrity.
  Interventions: Dietary Supplement: Golden Rice Cookies Without Piper Crocatum

INTERVENTIONS:
Dietary Supplement: Golden Rice Cookies With Piper Crocatum — This intervention consists of a functional food product in the form of cookies made from golden rice flour, enriched with Piper crocatum (red betel leaf extract). The cookies are administered orally, once daily, over a 28-day period. What distinguishes this intervention from others is the combination of golden rice a biofortified grain rich in beta-carotene with Piper crocatum, a traditional Indonesian medicinal plant known for its antioxidant and anti-inflammatory properties. The formulation is designed to target diabetic neuropathy prevention by enhancing neuroprotective effects through dietary supplementation. The product is standardized in dosage, appearance, and packaging to support double-blind administration and ensure consistency across participants.
  Arms: Golden Rice Cookies Enriched with Piper Crocatum
Dietary Supplement: Golden Rice Cookies Without Piper Crocatum — This intervention consists of cookies made from golden rice flour without the addition of Piper crocatum (red betel leaf extract). The cookies are administered orally, once daily, for 28 consecutive days. Although lacking the herbal component, golden rice itself is a biofortified grain rich in beta-carotene, offering nutritional value. The control product is matched in appearance, taste, and packaging to the experimental cookies to maintain double-blind conditions. This intervention serves as an active comparator to isolate the effect of Piper crocatum in preventing diabetic neuropathy symptoms
  Arms: Golden Rice Cookies Without Piper Crocatum

SUMMARY:
Diabetes mellitus is a chronic disease that can cause many complications, one of the most common being diabetic neuropathy. This condition occurs due to long-term high blood sugar levels that damage the nerves. Symptoms include tingling, burning, pain, and loss of sensation in the feet. If not prevented, neuropathy can progress to diabetic foot ulcers and even lead to amputation.

This study aims to evaluate whether Golden Rice Cookies enriched with Red Betel Leaf (Piper crocatum) can help prevent diabetic neuropathy in patients with diabetes. Golden rice is a type of rice that contains beta-carotene (provitamin A) and high fiber, which help maintain stable blood sugar levels and reduce oxidative stress. Meanwhile, red betel leaf contains flavonoids, polyphenols, and alkaloids with antioxidant, anti-inflammatory, and hypoglycemic properties that may protect nerves from damage.

Cookies were chosen as the intervention form because they are practical, easy to consume, and widely accepted by patients. In this study, patients will be divided into two groups: an intervention group receiving golden rice cookies with red betel leaf extract, and a control group receiving golden rice cookies without the extract. Changes in neuropathy symptoms will be assessed using the Neuropathy Symptom Score (NSS) before and after the intervention.

The expected outcome of this research is to provide scientific evidence that the combination of golden rice and red betel leaf in the form of cookies can serve as an effective, safe, and acceptable functional food to help prevent diabetic neuropathy. This nutritional intervention may support comprehensive diabetes management and improve patients' quality of life.

DETAILED DESCRIPTION:
Diabetes mellitus is a chronic metabolic disease with a steadily increasing prevalence worldwide. One of its most common and burdensome complications is diabetic neuropathy, which affects up to 50% of patients with type 2 diabetes. This condition is characterized by pain, tingling, or loss of sensation, particularly in the feet, and is a major risk factor for diabetic foot ulcers and amputations. Current management strategies mainly focus on strict glycemic control and the treatment of neuropathic pain, while preventive nutritional approaches remain limited.

With the growing interest in functional foods, new opportunities have emerged to support diabetes care. Golden rice, genetically enriched with beta-carotene (provitamin A), provides antioxidant and anti-inflammatory benefits along with dietary fiber that helps stabilize blood glucose levels. Red betel leaf (Piper crocatum), traditionally used in herbal medicine, contains flavonoids, polyphenols, and alkaloids with antioxidant, anti-inflammatory, and hypoglycemic properties that may protect nerves from damage caused by chronic hyperglycemia. The combination of these two functional ingredients offers promising neuroprotective potential for the prevention of diabetic neuropathy.

This study is designed as a randomized controlled trial using cookies made from golden rice enriched with Piper crocatum as the intervention. Cookies are chosen as the delivery form because they are practical, well-accepted by patients, and easy to consume regularly compared with supplements or herbal preparations. Participants will be divided into two groups: an intervention group receiving golden rice cookies with Piper crocatum extract, and a control group receiving golden rice cookies without the extract.

Throughout the 28-day intervention period, changes in neuropathy symptoms will be evaluated using the Neuropathy Symptom Score (NSS) before and after consumption. The study aims to determine whether the addition of Piper crocatum provides added benefits in preventing or reducing neuropathy symptoms compared with golden rice cookies alone.

This research is expected to provide scientific evidence on the role of combining golden rice and Piper crocatum in cookie form as an innovative functional food for the prevention of diabetic neuropathy. Such a nutritional intervention may offer an effective, safe, affordable, and acceptable strategy to support comprehensive diabetes management and improve patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 59 years
* Diagnosed with diabetes mellitus based on medical records
* Able to read and communicate effectively
* Willing to participate in the study, sign the informed consent form, and commit to consuming the cookies according to the prescribed dosage

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients with a history of allergy to any component of the intervention, including golden rice or Piper crocatum
* Patients with active diabetic foot ulcers

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Neuropathy Symptoms Score (NSS) | Baseline (Day 0) to Day 28
  Neuropathy Symptoms Score (NSS) is a standardized questionnaire used to assess the severity of peripheral neuropathy symptoms in patients with diabetes. The instrument evaluates common neuropathic symptoms including numbness, burning sensation, tingling, cramps, and pain. Each symptom is scored based on presence and characteristics (e.g., location, timing, aggravating factors), with a total score ranging from 0 to 9, where higher scores indicate more severe neuropathic symptoms. Assessment is conducted through participant interview by trained clinical assessors

SECONDARY OUTCOMES:
Fasting Blood Glucose Level | Baseline Day 0, Day 14, and Day 28
  Fasting blood glucose is measured using a point-of-care glucometer (IVD brand), following standard capillary blood sampling procedures. Participants undergo at least 8 hours of overnight fasting before measurement. A finger-prick capillary blood sample is applied to a compatible test strip, and the glucometer automatically analyzes and displays glucose concentration in mg/dL. Higher values indicate poorer glycemic control. All measurements are performed by trained research staff using calibrated devices according to the manufacturer's instructions.
Change in Peripheral Sensation Via Monofilament Test | Baseline (Day 0) and Post intervention (Day 28)
  Peripheral sensory response will be evaluated using the 10-gram Semmes-Weinstein monofilament test in diabetic patients without clinically diagnosed neuropathy. The test assesses protective sensation in the feet. Improvement or stabilization of sensory response after intervention indicates a potential preventive effect against diabetic neuropathy

OTHER OUTCOMES:
Adherence to Cookie Consumption | Daily from Day 1 to Day 28
  Adherence will be assessed using a daily consumption log provided to each participant. The log records whether the cookie was consumed each day from Day 1 to Day 28, along with any complaints or side effects experienced. Compliance will be calculated as the percentage of days the cookie was consumed as instructed. This measure also allows qualitative monitoring of tolerability and participant-reported issues during the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Andina Setyawati, S.Kep.,Ns.,M.Kep, Study Director — Faculty of Nursing, Hasanuddin University
Locations (1):
- UPTD Puskesmas Lompeta Singgani Tambu, Donggala, Central Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to confidentiality concerns and limited data management resources. The study is conducted in a primary care setting with restricted infrastructure for secure data sharing. All data will be used solely for internal analysis and reporting purposes.

REFERENCES:
- [Background] Setyawati A, Saleh A, Tahir T, Yusuf S, Syahrul S, Aminuddin A, Raihan M, Jafar N, Hamzah H, Arfian N. Matrix Metalloproteinase-9 Testing of Golden Rice Cookies With Piper Crocatum Active Extract for Preventing Foot Ulcers in Patients With Diabetes: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Feb 29;13:e49940. doi: 10.2196/49940. PMID 38422498
- [Result] Dyck PJ, Kratz KM, Karnes JL, et al. The Neuropathy Symptom Score: A systematic measure for evaluation of distal symmetric polyneuropathy in clinical research. Neurology. 1997;48(3):593-601.
- [Result] Setyawati A, Wahyuningsih MSH, Nugrahaningsih DAA, Effendy C, Fneish F, Fortwengel G. Piper crocatum Ruiz & Pav. ameliorates wound healing through p53, E-cadherin and SOD1 pathways on wounded hyperglycemia fibroblasts. Saudi J Biol Sci. 2021 Dec;28(12):7257-7268. doi: 10.1016/j.sjbs.2021.08.039. Epub 2021 Aug 19. PMID 34867030
- See also: Official Website of The Faculcy of Nursing, Hasanuddin University — https://nursing.unhas.ac.id/
- See also: Hasanuddin University Official Website — https://unhas.ac.id/